CLINICAL TRIAL: NCT01452815
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Evaluation of the Efficacy and Safety of Once-Daily Administrations of TZP-102 for the Treatment of Symptoms Associated With Diabetic Gastroparesis
Brief Title: Affects of Once-daily Oral Administration of TZP-102 on the Treatment of Symptoms Associated With Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tranzyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TZP-102-CL-G003
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2012-08

CONDITIONS: Gastroparesis; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: diabetic gastroparesis; delayed gastric emptying; gastroparesis; diabetes mellitus, Type 1; diabetes mellitus, Type 2
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Drug: placebo
  Interventions: Drug: Placebo
- 2 (Experimental): 10mg TZP-102
  Interventions: Drug: 10mg TZP-102
- 3 (Experimental): 20mg TZP-102
  Interventions: Drug: 20mg TZP-102

INTERVENTIONS:
Drug: Placebo — Two #2 oval shaped,opaque-white, hard gelatin shell capsules containing inactive ingredients taken orally once daily for 12 weeks.
  Arms: 1
Drug: 10mg TZP-102 — One 10mg #2 oval shaped, opaque-white, hard gelatin shell capsule containing active ingredients and one placebo capsule each taken orally once daily for 12 Weeks
  Arms: 2
Drug: 20mg TZP-102 — Two 10mg #2 oval shaped, opaque-white, hard gelatin shell capsules containing active ingredients
  Arms: 3

SUMMARY:
The purpose of this study is to test the safety and effectiveness of two dosage levels (10mg and 20mg) of TZP-102 compared to placebo (capsule that looks like the study drug but contains no active drug), administered once-daily for 12 weeks, in diabetic subjects with symptoms associated with gastroparesis.

DETAILED DESCRIPTION:
Considered subjects will be screened to determine eligibility for entry into the study. The Screening Visit must take place at least 14 days, but not more than 21 days, before the planned date of study entry (randomization and administration of the first dose of study drug on Study Day 1). The baseline evaluation of gastric emptying must be scheduled at least 7 days (in the U.S.) and 10 days (in Europe) before the Day 1 Visit. Subjects will answer questions relating to their gastroparesis symptoms in an electronic diary (like a palm pilot) beginning on the first day of the screening period.

Eligible subjects will be randomized to receive placebo or one of two dosages of TZP-102 (10mg or 20mg) once daily for 12 weeks. After randomization and administration of the first dose of study drug on Study Day 1 (the Study Entry Visit), subsequent visits to the clinic will be scheduled every two weeks during the 12-week Treatment period and 4-week Follow-Up Period.

All visits will be conducted on an outpatient basis. Visits for a given subject throughout the study should be scheduled to start at approximately the same time, in the morning. Subjects will be instructed to take their daily dose of study drug each morning (when not attending a study visit), at least 30 minutes before breakfast. Subjects will be instructed to not take study drug on the morning of each treatment period visit and to bring study drug supplies with them to the clinic; study drug will be administered in the clinic after all scheduled assessments/procedures (after all pre-dose assessments at each of the Day 1 and Week 12 Visits) are completed.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age, inclusive
* Type 1 or type 2 diabetes mellitus
* History of symptoms of gastroparesis for at least 3 months leading up to the Screening Visit
* Gastric half-emptying time >82 minutes, demonstrated by the Gastric Emptying Breath Test performed at the Screening Visit OR documented delayed gastric emptying within the previous 24 months
* Mild to moderate severity of gastroparesis symptoms during the screening period
* Body Mass Index (BMI) < 45.0 at the Screening Visit
* Glycosylated hemoglobin (HbA1c) level < 11.0% at the Screening Visit
* Upper gastrointestinal obstruction ruled out by endoscopy or barium scan
* Concomitant medications must be stable for at least 2 weeks leading up to the Baseline Visit and must be maintained during the study.
* Females of child-bearing potential must have a negative serum pregnancy test and use (and agree to continue to use throughout the study) an acceptable form of contraception.

Exclusion Criteria:

* Persistent daily vomiting
* Gastrectomy, bariatric surgery, fundoplication or vagotomy/pyloroplasty
* Has had or plans to have endoscopic pyloric injections of botulinum toxin within 6 months prior to the Screening Visit or during the study.
* NG, PEG or PEJ feeding tube within 2 weeks prior to the Screening Visit
* Required in-patient hospitalization for treatment of gastroparesis within 2 weeks prior to the Screening Visit
* Required parenteral nutrition for treatment of gastroparesis within 2 months prior to the Screening Visit
* Active gastric pacemaker within 3 months prior to the Screening Visit
* Participated in an investigational study within 30 days prior to the Screening Visit
* Chronic severe diarrhea
* Diabetic ketoacidosis that required inpatient hospitalization within 30 days prior to the Screening Visit
* History of any eating disorder within 2 years prior to the Screening Visit
* Chronic obstructive pulmonary disease (COPD) or chronic asthma
* Chronic smoker that is unable or unwilling to abstain from smoking during the two visits that the gastric emptying breath test will be performed
* History of risk factors for Torsades de Pointes
* Corrected QT interval calculated using Fredericia's formula >= 500 msec, recorded and confirmed on any of the three ECG assessments performed during the screening period
* Bradycardia or hypotension assessed as clinically-significant by the investigator
* Requires treatment with concomitant medication that is a substrate of Cytochrome P450 isoenzyme 3A4 and known to have a clinically recognized risk for Torsades de Pointes
* History of acute myocardial infarction, unstable angina or a transient (cerebral) ischemic attack within 12 months prior to the Screening Visit
* History of severe depression, psychiatric disorder or cognitive impairment
* History of alcohol or drug abuse or dependency within 2 years prior to the Screening Visit
* Taking opiates for abdominal pain
* Known history of Hepatitis B or C or HIV infection
* Requires dialysis or elevated creatinine at the Screening Visit
* Abnormal liver function tests at the Screening Visit
* Uncontrolled hypo- or hyperthyroidism
* Adrenal insufficiency
* Active malignancy other than basal cell or squamous cell carcinoma of the skin
* Pregnant or breast-feeding
* Allergies to components of the breath test meal or severe lactose intolerance
* Any other medical condition or social circumstance that, in the investigator's opinion, makes it inappropriate for the patient to participate in this clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in symptoms associated with diabetic gastroparesis | 12 Weeks

SECONDARY OUTCOMES:
Change from baseline on health-related quality of life | 12 Weeks
Adverse Events (AEs) | 12 Weeks
Cardiovascular Parameters (blood pressure, heart rate, 12-Lead ECG) | 12 Weeks
Clinical Chemistry and Hematology Parameters | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Connie Cosentino, Study Director — Tranzyme Pharma
Locations (51):
- United States (30):
  - Tranzyme Investigational Site, Huntsville, Alabama
  - Tranzyme Investigational Site, Tucson, Arizona
  - Tranzyme Investigational Site, Jonesboro, Arkansas
  - Tranzyme Investigational Site, Little Rock, Arkansas
  - Tranzyme Investigational Site, Long Beach, California
  - Tranzyme Investigational Site, Stanford, California
  - Tranzyme Investigational Site, Ventura, California
  - Tranzyme Investigational Site, Hialeah, Florida
  - Tranzyme Investigational Site, Inverness, Florida
  - Tranzyme Investigational Site, Jacksonville, Florida
  - Tranzyme Investigational Site, Miami, Florida
  - Tranzyme Investigational Site, New Smyrna Beach, Florida
  - Tranzyme Investigational Site, Port Orange, Florida
  - Tranzyme Investigational Site, Oak Lawn, Illinois
  - Tranzyme Investigational Site, Anderson, Indiana
  - Tranzyme Investigational Site, Kansas City, Kansas
  - Tranzyme Investigational Site, Monroe, Louisiana
  - Tranzyme Investigational Site, Boston, Massachusetts
  - Tranzyme Investigational Site, Mexico, Missouri
  - Tranzyme Investigational Site, Fayetteville, North Carolina
  - Tranzyme Investigational Site, Raleigh, North Carolina
  - Tranzyme Investigational Site, Salisbury, North Carolina
  - Tranzyme Investigational Site, Winston-Salem, North Carolina
  - Tranzyme Investigational Site, Oklahoma City, Oklahoma
  - Tranzyme Investigational Site, Portland, Oregon
  - Tranzyme Investigational Site, Philadelphia, Pennsylvania
  - Tranzyme Investigational Site, Jackson, Tennessee
  - Tranzyme Investigational Site, El Paso, Texas
  - Tranzyme Investigational Site, Houston, Texas
  - Tranzyme Investigational Site, Tacoma, Washington
- Belgium (3):
  - Tranzyme Investigational Site, Bruges
  - Tranzyme Investigational Site, Brussels
  - Tranzyme Investigational Site, Ghent
- Denmark (3):
  - Tranzyme Investigational Site, Aarhus
  - Tranzyme Investigational Site, Gentofte Municipality
  - Tranzyme Investigational Site, Odense
- Finland (2):
  - Tranzyme Investigational Site, Porvoo
  - Tranzyme Investigational Site, Tampere
- Germany (3):
  - Tranzyme Investigational Site, Essen
  - Tranzyme Investigational Site, Mainz
  - Tranzyme Investigational Site, Stuttgart
- Tranzyme Investigational Site, Bergen, Norway
- Poland (7):
  - Tranzyme Investigational Site, Bialystok
  - Tranzyme Investigational Site, Bydgoszcz
  - Tranzyme Investigational Site, Kielce
  - Tranzyme Investigational Site, Krakow
  - Tranzyme Investigational Site, Lodz
  - Tranzyme Investigational Site, Olsztyn
  - Tranzyme Investigational Site, Warsaw
- Sweden (2):
  - Tranzyme Investigational Site, Stockholm
  - Tranzyme Investigational Site, Uppsala

REFERENCES:
- [Derived] McCallum RW, Lembo A, Esfandyari T, Bhandari BR, Ejskjaer N, Cosentino C, Helton N, Mondou E, Quinn J, Rousseau F; TZP-102 Phase 2b Study Group. Phase 2b, randomized, double-blind 12-week studies of TZP-102, a ghrelin receptor agonist for diabetic gastroparesis. Neurogastroenterol Motil. 2013 Nov;25(11):e705-17. doi: 10.1111/nmo.12184. Epub 2013 Jul 15. PMID 23848826